CLINICAL TRIAL: NCT05244642
Title: A Randomized, Open, Multi-center Phase III Study to Evaluate the Efficacy and Safety of Penpulimab Monotherapy vs. Standard Chemotherapy Selected by Investigator in the Relapsed and Refractory Classical Hodgkin's Lymphoma (R/R cHL)
Brief Title: A Phase III Study to Evaluate the Efficacy and Safety of Penpulimab in the Relapsed and Refractory Classical Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK105-303
Record Dates: First submitted 2022-01-25; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Hodgkin Disease Lymphoma
MeSH Terms: interventions — penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Penpulimab) (Experimental): Participants receive Penpulimab 200mg intravenously (IV) on Day 1, Q2W for 24 months.
  Interventions: Drug: Penpulimab
- Group B (Chemotherapy) (Active Comparator): Participants receive investigator's choice of chemotherapy Q2W or Q3W for up to 4 or 6 cycles.
  Interventions: Drug: Investigator's choice of Chemotherapy

INTERVENTIONS:
Drug: Penpulimab — A humanized monoclonal immunoglobulin.
  Other Names: AK105
  Arms: Group A (Penpulimab)
Drug: Investigator's choice of Chemotherapy — Participants will receive one of the following chemotherapies, including but not limited to DHAP (cisplatin 100mg/m2 D1, high dose cytarabine 2 mg/m2 q12h D2, dexamethasone 40mg D1-4, Q3W); ESHAP (etoposide 40 mg/m2 D1-4, cisplatin 25 mg/m2 D1-4, high dose cytarabine 2 mg/m2 D5, methylprednisolone 500mg D1-4, Q3W); DICE (dexamethasone 10mg/m2 D1-4, ifosfamide 1.0g/m2 D1-4, cisplatin 25mg/m2 D1-4, etoposide 60 mg/m2 D1-4, Q3W); ICE (ifosfamide 5 mg/m2 D2, carboplatin AUC 5 D2, etoposide 100 mg/m2 D1-3, Q3W); IGEV (ifosfamide 2 mg/m2 D1-4, gemcitabine 800 mg/m2 D1, D4, vinorelbine 20mg/m2 D1, prednisone 100 mg D1-4, Q3W); GVD (gemcitabine 1g/m2 D1, D8, vinorelbine 20 mg/m2 D1, D8, liposome doxorubicin 15 mg/m2 D1, D8, Q3W); MINE (etoposide 65mg/m2 D1-3, ifosfamide 1.33g/m2 D1-3, mitoxantrone 8mg/m2 d1, Q3W); GemOx (gemcitabine 800mg/m2 D1, D8, oxaliplatin 85mg/m2 D1, Q3W); GemOx (gemcitabine 1000mg/m2 D1, oxaliplatin 100mg/m2d1, Q2W).
  Arms: Group B (Chemotherapy)

SUMMARY:
This is an open-label, multicenter, randomized, phase 3 trial to evaluate the efficacy of Penpulimab vs. standard chemotherapy selected by investigator in patients with relapsed or refractory classic Hodgkin's lymphoma.

DETAILED DESCRIPTION:
This is an open-label, multicenter, randomized, phase 3 trial to evaluate the efficacy of Penpulimab in patients with relapsed or refractory classic Hodgkin's lymphoma. Participants will be randomized to receive either Penpulimab monotherapy or chemotherapy of investigators' choice. The primary hypotheses of this study are that treatment with Penpulimab prolongs Progression-free Survival (PFS) in participants with relapsed or refractory Classical Hodgkin Lymphoma compared to treatment with Chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent form (ICF).
2. Age of ≥ 18 years at the time of enrollment, male or female.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy of ≥ 3 months.
5. Histologically confirmed classic Hodgkin's lymphoma (cHL).
6. Relapsed (disease progression during or after most recent therapy) or refractory (failure to achieve CR or PR after most recent therapy) cHL and meet any of the following criterions:

   1. Subjects who have received autologous hematopoietic stem cell transplantation (ASCT) after salvage chemotherapy, followed by relapse or progression.
   2. For subjects who have not received ASCT, it is required at least 2 lines of prior systemic chemotherapy. Refractory subjects are defined as failure to achieve PR after at least 2 cycles of chemotherapy, or failure to achieve CR after at least 4 cycles of chemotherapy. If the best response to treatment is PD or the reason for ending the treatment is PD, the subject is considered as refractory without requirement on the number of cycles of treatment received.
7. Have at least one measurable lesion according to Lugano classification 2014.
8. Have adequate hematologic and organ function as defined below:

   1. Hematology (supportive treatment with ang blood components or cell growth factors is not allowed within 7 days prior to enrollment laboratory test): Absolute neutrophil count (ANC) ≥ 1.0x109/L, platelet count ≥ 75 x109/L, hemoglobin ≥ 80g/L.
   2. Kidney: Serum creatinine ≤ 1.5 X ULN and estimated GFR (by Cockroft-Gault equation) ≥ 50ml/min.
   3. Liver: Total bilirubin ≤ 1.5 X ULN, AST/ALT ≤ 2.5 X ULN.
   4. Coagulation: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
9. Women of childbearing potential (WOCBP) must be tested for serum or urine pregnancy negative within 3 days prior to the first dose of study treatment. WOCBP will be instructed to adhere to contraception while on treatment and for at least 150 days after the last dose of study treatment. Male subjects who are sexually active with WOCBP will be instructed to adhere to contraception while on treatment and for at least 150 days after receiving the last dose of study treatment.

Exclusion Criteria:

1. Nodular lymphocytes are non-Hodgkin's lymphoma or gray area lymphoma.
2. Central nervous system lymphoma invasion.
3. Have received any investigational treatment or investigational device within 4 weeks prior to the first dose of study treatment.
4. Enrolled in another clinical study at the same time, unless it is an observational (non-interventional) clinical study or in follow-up period for interventional studies.
5. The last radiotherapy or last anti-tumor therapy (chemotherapy, tumor embolization, etc.) has been given within 4 weeks prior to the first dose of study treatment.
6. Prior exposure to any anti-PD-1, anti-PD-L1, anti-CTLA-4 antibody, or any other antibody or drug target for T cell co-stimulatory or checkpoint pathways, such as ICOS or agonists (e.g., CD40, CD137, GITR and OX40, etc.).
7. Subjects with other malignancy within 5 years prior to the first dose of study treatment, except for locally curable cancers that have been apparently cured, such as basal or skin squamous cell carcinoma, superficial bladder cancer, cervix or breast carcinoma in situ.
8. Active, known or suspected autoimmune disease, or medical history of autoimmune disease in the past 2 years, with the exceptions of vitiligo, alopecia, graves' disease, psoriasis or eczema not requiring systemic treatment within the last 2 years, asymptomatic but only steady doses of hormone replacement therapy are required for hypothyroidism (caused by autoimmune thyroiditis) or type I diabetes requiring only a steady dose of insulin replacement therapy, or that the primary disease does not relapse without external triggering factors
9. Systemic glucocorticoids or other immunosuppressive drugs used within 7 days prior to the first dose of study treatment. It is allowed to use nasal spray, inhaled, or other topical application of glucocorticoids, and a physiological dose of systemic glucocorticoids does not exceed 10 mg/ day or the equivalent. Glucocorticoids are also allowed to temporary use for the treatment of dyspnea symptoms of chronic obstructive pulmonary disease (COPD), or as a prophylactic agent for hypersensitivity reactions.
10. Known active human immunodeficiency virus (HIV) positive.
11. Known history of primary immunodeficiency.
12. Known active tuberculosis.
13. Prior solid organ transplantation, allogeneic hematopoietic stem cell transplantation (HSCT).
14. ASCT within 90 days prior to the first dose of study treatment.
15. History of gastrointestinal perforation and/ or fistula (patients can be enrolled if the gastrointestinal perforation or fistula has been surgically removed), ileus (including incomplete ileus requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection with chronic diarrhea), Crohn's disease, ulcerative colitis or chronic diarrhea within 6 months prior to the first dose of study treatment.
16. Known history of or active interstitial lung disease (ILD) or ILD needs to use corticosteroids.
17. Patients with untreated chronic hepatitis B virus (HBV) infection or chronic HBV carriers with HBV DNA exceeding 500 IU/ mL, or hepatitis C virus (HCV) infection. Patients with non-active HBsAg carriers, treated and stable (HBV DNA <500 IU/ mL), and cured HCV infection can be enrolled. Patients with HCV seropositivity are eligible only if the HCV RNA test negative.
18. Major surgery (craniotomy, thoracotomy, or laparotomy) performed within 30 days prior to the first dose of study treatment, or not fully recovered from previous surgery. Local procedures (such as systemic placement of ports, prostate biopsy) are allowed, provided that which are completed at least 24 hours prior to the first dose of study treatment.
19. Subjects with uncontrolled pleural effusion or ascites.
20. Active infection requiring systemic treatment.
21. Uncontrolled concurrent conditions, including but not limited to persistent or active infection, symptomatic congestive heart failure (NYHA grade 3 or 4), uncontrolled hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg), unstable angina, arrhythmia, or other mental illness/social conditions may limit the subject's compliance with the study requirements or impair the ability of the subject to provide written informed consent.
22. Known history of arterial or venous thrombosis events within 6 months prior to the first dose of study treatment, including myocardial infarction, unstable angina, and cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or any other severe thromboembolism. Except for infusion port or catheter-derived thrombosis, or superficial venous thrombosis, or thrombosis that keep stable after conventional anticoagulant therapy.
23. Unresolved toxicities from prior anti-tumor treatment, defined as toxicity that has not recovered to NCI CTCAE V5.0 Grade 0 or 1, or to levels specified in inclusion/ exclusion criteria, except for alopecia. Subjects with irreversible toxicity that will not worsen after administration of study drugs as evaluated by investigator (e.g., hearing loss) may be eligible after discussion with Sponsor.
24. Have received live or attenuated vaccine(s) within 30 days prior to the first dose of study treatment, or plan to receive live or attenuated vaccine(s) during the study.
25. Known allergy to any components or any ingredients of penpulimab and chemotherapy agents selected by investigator.
26. Pregnant or lactating women.
27. Subjects with NCI CTCAE v5.0 Grade ≥2 peripheral neuropathy.
28. Any conditions that evaluated by investigator may affect subjects' safety, or may interfere with the evaluation of study drug, or may confound the interpretation of study results.
29. Uncontrolled metabolic disorders, local or systemic manifestations either due to concomitant disease or the primary tumor, with high risk and/or uncertainty in survival evaluation, such as tumor leukemoid reaction (white blood cell count > 20×109/L), cachexia (known weight loss of more than 10% in the 3 months before screening), etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) assessed by Independent Radiologic Review Committee (IRRC) per Lugano Classification 2014 | Up to 2 years
  Time from the date of randomization to the date of progressive disease (PD) or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to end of study
  Time from the date randomization to death from any cause.
Objective Response Rate (ORR) | Up to 2 years
  ORR defined as the proportion of subjects who achieves a best overall response of CR or PR based on Lugano 2014 classification.
Disease Control Rate (DCR) | Up to 2 years
  DCR defined as the proportion of subjects' response of CR, PR, or SD based on Lugano Classification 2014.
Duration of Response (DoR) | Up to 2 years
  DoR defined as the time from the date that CR or PR are first occurred to the date of objective disease progression or death, whichever occurs first.
Time to Response (TTR) | Up to 2 years
  TTR defined as the time from the date of randomization to the date when the response criteria are first met, based on Lugano Classification 2014.
Number of subjects with adverse events (AEs) | From the time of signed informed consent through 90 days after the last dose of penpulimab
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment
Anti-drug antibody (ADA) | From first dose of penpulimab through to 30 days after last dose of penpulimab
  Number of subjects with detectable anti-drug antibody (ADA).

CONTACTS AND LOCATIONS:
Overall Officials: Yuqin Song, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (6):
- China (6):
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Beijing Cancer Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No